CLINICAL TRIAL: NCT01721811
Title: Retinal Function in Relation to Transient or Chronic Challenges to Retinal Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Oliver Niels Klefter, MD, Glostrup University Hospital, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Klefter2
Record Dates: First submitted 2012-10-31; First posted 2012-11-06 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Individuals; Patients With Diabetes.
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy (Experimental): Healthy study participanats
  Interventions: Other: Hyperoxia; Other: Glucose
- Diabetes (Experimental): Patients with diabetes
  Interventions: Other: Hyperoxia; Other: Glucose

INTERVENTIONS:
Other: Hyperoxia
  Other Names: Hyperoxia is achieved by short-term pure oxygen breathing.
Other: Glucose
  Other Names: Standardised oral glucose load.

SUMMARY:
The aim of the study is to investigate how the retina adapts to different metabolic challenges, e.g. chronic systemic hypoxia, hyperglycemia, special training conditions or diets as well as transient changes in the content of oxygen and glucose in the blood.

ELIGIBILITY:
Healthy individuals

Inclusion Criteria:

* Healthy volunteers.
* No known systemic or ocular disease.

Exclusion Criteria:

* Any systemic or ocular disease.

Patients with diabetes

Inclusion criteria:

* Diabetes mellitus
* No intraocular disease other than conditions attributable to diabetes.

Exclusion criteria:

* Intraocular disease other than conditions attributable to diabetes.
* Systemic conditions which might contraindicate hyperoxic stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Retinal vessel diameters during hyperoxia | Before hyperoxia, after 15 minutes of hyperoxia, 30 minutes after ending hyperoxia
  Measurement of retinal vessel diameters before, during and after hyperoxic stimulation.
Retinal perfusion velocities during hyperoxia | Before hyperoxia, after 15 minutes of hyperoxia, 30 minutes after ending hyperoxia
  Measurement of retinal perfusion velocities before, during and after hyperoxic stimulation.
Retinal oximetry during hyperoxia | Before hyperoxia, after 15 minutes of hyperoxia, 30 minutes after ending hyperoxia
  Measurement of retinal oximetry status before, during and after hyperoxic stimulation.
Retinal vessel diameters during hyperglycemia | Before glucose ingestion, every 30 minutes for 3 hours following oral glucose load
  Measurement of retinal vessel diameters before, during and after hyperglycemic stimulation.
Retinal perfusion during hyperglycemia | Before glucose ingestion, every 30 minutes for 3 hours following oral glucose load
  Measurement of retinal perfusion velocities before, during and after hyperglycemic stimulation.
Retinal oximetry during hyperglycemia | Before glucose ingestion, every 30 minutes for 3 hours following oral glucose load
  Measurement of retinal oximetry status before, during and after hyperglycemic stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klefter, MD, Principal Investigator — Glostrup UH; Michael Larsen, Professor, DMSci, Study Director — Glostrup UH
Locations (1):
- Department of Ophthalmology, Glostrup University Hospital, Glostrup Municipality, Denmark